CLINICAL TRIAL: NCT00115466
Title: Phase II Clinical Trial, Multicentre, Randomised and Comparative, to Evaluate the Efficacy and Safety of a New Therapy With Autologous Stem Cells Derived From Lipoaspirates for the Non-Surgical Treatment of Complex Perianal Fistula
Brief Title: Autologous Stem Cells Derived From Lipoaspirates for the Non-Surgical Treatment of Complex Perianal Fistula
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cellerix (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX401/TCFIS; Nr. 04-0211
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Anal Fistula
Keywords: ASCs (adult stem cells derived from adipose tissue); Fistula; Cell Therapy; Complex perianal fistula
MeSH Terms: conditions — Rectal Fistula; Fistula

INTERVENTIONS:
Procedure: Non-surgical autologous implant of ASCs

SUMMARY:
This comparative, multicentre, randomised clinical trial is designed with two parallel groups that will follow a treatment either with an autologous implant of ASCs (Adipose Derived Stem Cells) and fibrin glue (tissue adhesive material) or with fibrin glue alone for the non-surgical treatment of complex perianal fistula.

DETAILED DESCRIPTION:
Comparative, multicentre, randomised clinical trial, designed with two parallel groups that will follow a treatment either with an autologous implant of ASCs (Adipose Derived Stem Cells) and fibrin glue (tissue adhesive material) or with fibrin glue alone for the NON-SURGICAL treatment of complex perianal fistula. The closure/healing of the fistula will be evaluated periodically, and it will be considered completely closed if there is no suppuration from the external orifice and re-epithelialisation can be observed at 8 weeks after the administration of the randomised therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes older than 18 years of age.
* Patients with a complex perianal fistula pathology which we define as the subjects that fulfil some of the following conditions:

  * No palpation of the fistula tract beneath the perianal skin.
  * A tract that is parallel to the rectum on exploration with a stylet.
  * Associated faecal incontinence.
  * Risk factors of anal incontinence.
  * At least one previous operation for a fistulous disorder.
  * Suprasphincteric trajectories
  * Rectovaginal fistula
  * Prior diagnosis of Crohn's disease.
* Patients from whom written informed consent has been obtained for them to participate in the study prior to performing any procedure described in the study.
* Patients that have already been subjected to a colonoscopy within a period of up to 6 months prior to the study.

Exclusion Criteria:

* Patients that are extremely thin who should not be subjected to liposuction.
* Known allergy to local anaesthetics or to bovine proteins
* History of neoplasia in the past 5 years.
* Patients with a diagnosis of active Tuberculosis at the moment of inclusion.
* Patients with prior positive markers for any of the following pathogens: Hepatitis B and C, HIV-1 or HIV-2.
* Any other medical condition that in the judgement of the investigator could interfere with their optimal participation in the study or produce a significant risk to the patient.
* Patients that have participated in another study in the 30 days prior to this one or that have planned to participate simultaneously in another study.
* Patients that have not given their informed consent to participate in this study.
* Psychiatric disorder or other factors that in the judgement of the investigator could complicate the participation of the patient in the study.
* Breast feeding, gestation or intention to become pregnant up to 6 months after finalising their participation in the study, or that are not using adequate methods of contraception during the same period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-10; Study Completion 2006-07

PRIMARY OUTCOMES:
Complete closure at week 8 (defined as no suppuration from the external orifice and re-epithelization)

SECONDARY OUTCOMES:
No fistula recurrence after 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Damian Garcia-Olmo, Prof., Principal Investigator — Cellerix
Locations (1):
- Cellerix Sl, Tres Cantos, Madrid, Spain

REFERENCES:
- [Result] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590